CLINICAL TRIAL: NCT05759468
Title: NAD Augmentation to Treat Diabetes Kidney Disease: A Randomized Controlled Trial
Brief Title: NAD Augmentation in Diabetes Kidney Disease
Acronym: DKD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Boston Medical Center (Other)
Responsible Party: Principal Investigator, Shalendar Bhasin, MD, Principal Investigator, Professor of Medicine, Harvard Medical School Director, Research Program in Men's Health: Aging and Metabolism Co-Director, BWH Center for Transgender Health Director, Boston Claude D. Pepper Older Americans Independence Center, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021P003702
Record Dates: First submitted 2023-01-09; First posted 2023-03-08 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Type2diabetes; Diabetic Kidney Disease
Keywords: diabetes; type 2 diabetes; kidney disease
MeSH Terms: conditions — Diabetic Nephropathies; Diabetes Mellitus; Diabetes Mellitus, Type 2; Kidney Diseases

STUDY DESIGN:
Intervention Model Description: This will be two center, randomized, double-blind, placebo-controlled, parallel group trial to determine whether βNMN, after its daily oral administration, is associated with a greater reduction in the UACR compared to placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study is double-blind in that the study participants and the study staff involved in outcomes assessments will be unaware of the intervention assignment. The randomization schedule will be masked from all study personnel except those specifically designated below.
  1. The unblinded study biostatistician
  2. The staff of the Investigational Drug Pharmacy Services.
  3. The DSMB, if requested
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Investigational Product - MIB 626 (Active Comparator): The MIB-626 will be a GMP-grade microcrystalline solid NMN mixed with inert excipients (including microcrystalline cellulose) and compressed into tablets at a dose strength of 500 mg per tablet, enabling administration of the 1,000 mg twice daily using two tablets taken twice daily.
  Interventions: Drug: Investigational Product - MIB 626
- Placebo (Placebo Comparator): Participants randomized to placebo will receive Matching placebo tablets will be provided by Metro International Biotech, LLC.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Investigational Product - MIB 626 — The eligible participants will be assigned to receive either NMN or placebo using concealed block randomization in a 1:1 ratio, stratified by sex (male, female), age (60 to 75, >75 years) and trial site. The randomization list will be generated by the unblinded biostatistician using the software R (www.r-project.org), and deployed in a secure, centralized web-based application accessible to study staff following confirmation of a participant's eligibility.
  Other Names: NMN
  Arms: Investigational Product - MIB 626
Drug: Placebo — Placebo - Participants randomized to placebo will receive Matching placebo tablets will be provided by Metro International Biotech, LLC.
  Other Names: Placebo for NMN
  Arms: Placebo

SUMMARY:
A phase 2a trial randomized, double-blind, placebo-controlled, parallel group trial to determine whether NMN administration improves DKD, as indicated by a significantly greater reduction in UACR compared with placebo administration. Eligible participants will be randomized to receive either 1000 mg NMN or placebo twice daily.

DETAILED DESCRIPTION:
This will be two centers, randomized, double-blind, placebo-controlled, parallel group trial to determine whether βNMN, after its daily oral administration, is associated with a greater reduction in the UACR compared to placebo.

The trial will enroll community-dwelling older adults, 60 years or older, with type 2 diabetes mellitus (T2DM) and urine albumin to creatinine excretion ratio > 100 mg/ g creatinine.

ELIGIBILITY:
Inclusion Criteria:

1. Has T2DM, as indicated by any of the following:

   1. Self-report of diabetes plus the use of a prescribed diabetes medication.
   2. ICD-10 code for diabetes plus current use of a diabetes medication in the electronic medical record.
   3. HbA1c >6.4%; or 2 fasting glucose > 125 mg/dL
2. Fasting morning UACR between 100 and 2,000 mg/g creatinine on two separate days
3. If UACR is > 300 mg/g creatinine, must be currently using an ACE inhibitor or an ARB
4. eGFR > 30 mL/ min / 1.73 m2
5. Hemoglobin A1c <9%
6. Able to speak English or Spanish
7. Willing and able to provide written informed consent
8. In addition, female participants must Not be pregnant and not planning to become pregnant over the next 6 months

Exclusion Criteria:

1. Fasting morning UACR > 2,000 mg/ g creatinine
2. Other laboratory abnormalities:

   1. Has AST or ALT > 3 times the upper limit of normal
   2. creatinine > 2.5 mg/dL
   3. Hematocrit < 0.34 or 0.50 L/L
3. A major adverse cardiovascular event in preceding 3 months
4. Participation in an investigational trial to evaluate pharmaceuticals or biologics within the past 3 months or 5 half-lives, whichever is shorter
5. Hypoglycemia unawareness or other medical conditions which could jeopardize participant's safety.
6. History of alcohol or substance use disorder or dependence (DSM 5 criteria) within the last 2 years.
7. Major depressive disorder, bipolar disorder, schizophrenia, or current psychotic symptoms or behavioral problems that could interfere with study procedures.
8. BMI > 42.5 kg/ m2

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-04-13 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is the change from baseline in UACR over the 6-month intervention period. | 6 months
  To determine whether treatment with a microcrystalline formulation of β nicotinamide mononucleotide (βNMN) in older adults with DKD improves urinary albumin to creatinine excretion ratio (UACR), compared to placebo.

SECONDARY OUTCOMES:
Assess the proportion of participants in the two study arms with 30% or greater reduction in UACR | 6 months
  In supportive analysis of the primary outcome, the investigator will compare the proportion of participants in the two study arms with 30% or greater reduction in UACR
Assess the change from baseline over the 6-month intervention period in biomarkers of kidney injury. | 6 month
  Compared to placebo treatment, NMN treatment of older adults with DKD will assess for improvements in biomarkers of kidney injury in association with DKD prognosis by measuring KIM-1 and STNFR1 combinedly.
Change from baseline in the levels of serum creatinine over 6-month intervention period | 6 month
  To determine whether NMN treatment is associated with change in serum creatinine from baseline to 24 weeks between the two study arms.
Change from baseline in the levels of cystine C over 6-month intervention period. | 6 month
  To determine whether NMN treatment is associated with change in cystatin C from baseline to 24 weeks between the two study arms.
To determine whether NMN treatment is associated with significantly greater improvement in muscle endurance. | 6 month
  Assess the change from baseline in muscle endurance by exercises (reps to failure) using Keiser Machines
Assess the change from baseline in performance-based measures of function. | 6 month
  To determine whether NMN treatment is associated with significantly greater improvement in performance based by using 6-minute walking distance measure of function.
To determine whether NMN alters the circulating biomarkers of aging that the geroscience experts have recommended. | 6 months
  Compared to placebo treatment, NMN treatment will be assessed to identify greater changes in the circulating biomarkers of aging. the biomarkers that will be assessed are IL6 and TNFalpha
Assess the change from baseline in the levels of NMN in the peripheral blood and in the PBMCs using a validated LC-MS/MS assay. | 6 months
  NMN treatment will be assessed to determine significant increases in blood levels of NAD and its metabolome during the 24-week intervention period. The increase in NAD levels are to be observed during the intervention period in NMN-treated subjects that will be sustained during the 12-week follow-up period (legacy effect).
Assess the change in measure of H1bac as a measure of glycemic control over the 6 months intervention period. | 6 months
  To determine the effect of NMN treatment on Hb1ac (expressed in mg/dL) in the body as a measure of glycemic control.
Assess the change in measure of fasting glucose as a measure of glycemic control over the 6 months intervention period. | 6 months
  To determine the effect of NMN treatment on fasting glucose in the body as a measure of glycemic control.

CONTACTS AND LOCATIONS:
Overall Officials: Shalender Bhasin, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared